CLINICAL TRIAL: NCT07128173
Title: The Effect of Incubator Covers on the Sleep-wake Cycles of Newborn Babies: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ayşe Belpınar, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YBozokU
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Preterm Infants; Sleep
Keywords: Newborn; incubator cover; sleep,; wakefulness
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomised controlled experimental study with single-blind methodology.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incubator Cover Group (Experimental): Neonatal information form was filled and consent was obtained. Actigraphy and 24-hour sleep duration were recorded before incubator cover application.
  The incubators were covered with incubator covers for 24 hours.24-hour sleep durations were recorded again by actigraphy.
  Interventions: Other: Incubator Cover Group
- Control Group (Experimental): Neonatal information form was filled and consent was obtained. Actigraphy and 24-hour sleep duration were recorded.No practice other than routine medical treatment follow-up and nursing care was performed.24-hour sleep durations were recorded again by actigraphy.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Incubator Cover Group — Incubator Cover Group: Neonatal information form was filled and consent was obtained.
  Actigraphy and 24-hour sleep duration were recorded before incubator cover application.The incubators were covered with incubator covers for 24 hours.24-hour sleep durations were recorded again by actigraphy.
  Arms: Incubator Cover Group
Other: Control Group — Control Group:Neonatal information form was filled and consent was obtained. Actigraphy and 24-hour sleep duration were recorded. No practice other than routine medical treatment follow-up and nursing care was performed.24-hour sleep durations were recorded again by actigraphy.
  Arms: Control Group

SUMMARY:
This study investigated the effect of incubator covers on sleep-wakefulness in premature infants.The study was conducted using a randomised controlled experimental design. The study population consisted of premature in the 30-37 gestational week range who were admitted to the NICU of a hospital located in the Central Anatolia Region. The sample comprised 64 premature infants, who were divided into an incubator cover group (n = 32) and a control group (n = 32). Data were collected using a neonatal follow-up form and actigraphy. The incubator cover group received a 24-hour covers application. The control group received routine nursing care without any additional interventions. Pre-test and post-test assessments were conducted in both groups, and the 24-hour sleep patterns of the newborns were evaluated using actigraphy.

DETAILED DESCRIPTION:
Objective: This study investigated the effect of incubator covers on sleep-wakefulness in premature infants.

Materials and Methods: The study was conducted using a randomised controlled experimental design. The study population consisted of premature in the 30-37 gestational week range who were admitted to the NICU of a hospital located in the Central Anatolia Region. The sample comprised 64 premature infants, who were divided into an incubator cover group (n = 32) and a control group (n = 32). Data were collected using a neonatal follow-up form and actigraphy. The incubator cover group received a 24-hour covers application. The control group received routine nursing care without any additional interventions. Pre-test and post-test assessments were conducted in both groups, and the 24-hour sleep patterns of the newborns were evaluated using actigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Newborn babies in the Neonatal Intensive Care Unit who were born at 30-37 weeks of gestation.
* A birth weight of 1500 grams or more. Stable vital signs
* Corrected gestational age of 30-37 weeks (plus 7-10 days). Those between 7 and 10 days old

Exclusion Criteria:

* Those requiring high-frequency mechanical ventilation.
* Those receiving sedative treatment.
* Those with hyperbilirubinemia
* Infants with hypoglycaemia or hyperglycaemia

Ages: 30 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency (pre-test) | Actigraphy and 24-hour sleep duration were recorded before incubator cover application (pre-test)
  sleep parametres
Sleep duration minutes (pre-test) | 24-hour sleep durations were recorded again by actigraphy (pre-test)
  sleep parametres
Number of awakenings of the infant during sleep (pre-test) | Actigraphy and 24-hour sleep duration were recorded before incubator cover application (pre-test)
  sleep parametres
Wakefulness time minutes (pre-test) | Actigraphy and 24-hour sleep duration were recorded before incubator cover application (pre-test)
  sleep parametres
Sleep efficiency (post-test) | Actigraphy and 24-hour sleep duration were recorded before incubator cover application (post-test)
  sleep parametres
Sleep duration minutes (post-test) | Actigraphy and 24-hour sleep duration were recorded before incubator cover application (post-test)
  sleep parametres
Number of awakenings of the infant during sleep (post-test) | Actigraphy and 24-hour sleep duration were recorded before incubator cover application (post-test)
  sleep parametres
Wakefulness time minutes (post-test) | Actigraphy and 24-hour sleep duration were recorded before incubator cover application (post-test)
  sleep parametres

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Belpınar, pHD, Principal Investigator — Bozok University
Locations (1):
- Yozgat Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kok EY, Kaur S, Mohd Shukri NH, Abdul Razak N, Takahashi M, Teoh SC, Tay JEF, Shibata S. The role of light exposure in infant circadian rhythm establishment: A scoping review perspective. Eur J Pediatr. 2024 Dec 30;184(1):112. doi: 10.1007/s00431-024-05951-3. PMID 39738921
- [Background] Kuhn P, Zores C, Langlet C, Escande B, Astruc D, Dufour A. Moderate acoustic changes can disrupt the sleep of very preterm infants in their incubators. Acta Paediatr. 2013 Oct;102(10):949-54. doi: 10.1111/apa.12330. Epub 2013 Jul 19. PMID 23800026
- [Background] Lewis P, Wild U, Pillow JJ, Foster RG, Erren TC. A systematic review of chronobiology for neonatal care units: What we know and what we should consider. Sleep Med Rev. 2024 Feb;73:101872. doi: 10.1016/j.smrv.2023.101872. Epub 2023 Nov 8. PMID 38000120
- [Background] Neukamm AC, Quante M, Poets CF, Shellhaas RA; "Neonatal Sleep Talks (NEST)" group. The impact of sleep in high-risk infants. Pediatr Res. 2025 Dec;98(6):2073-2081. doi: 10.1038/s41390-025-04049-2. Epub 2025 Apr 10. PMID 40210954
- [Background] Orsi KC, Avena MJ, Lurdes de Cacia Pradella-Hallinan M, da Luz Goncalves Pedreira M, Tsunemi MH, Machado Avelar AF, Pinheiro EM. Effects of Handling and Environment on Preterm Newborns Sleeping in Incubators. J Obstet Gynecol Neonatal Nurs. 2017 Mar-Apr;46(2):238-247. doi: 10.1016/j.jogn.2016.09.005. Epub 2017 Jan 3. PMID 28056335
- [Background] Zores C, Dufour A, Pebayle T, Dahan I, Astruc D, Kuhn P. Observational study found that even small variations in light can wake up very preterm infants in a neonatal intensive care unit. Acta Paediatr. 2018 Jul;107(7):1191-1197. doi: 10.1111/apa.14261. Epub 2018 Feb 27. PMID 29412484